CLINICAL TRIAL: NCT01166139
Title: Phase IIA Study of the Safety and Tolerability of the Use of Nilotinib in the Treatment of Systemic Sclerosis
Brief Title: Nilotinib in the Treatment of Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Rudolph Rupert Scleroderma Program (Unknown); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10041
Record Dates: First submitted 2010-07-01; First posted 2010-07-20 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Systemic Sclerosis
Keywords: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib 400 mg twice daily (Experimental)
  Interventions: Drug: Nilotinib (Tasigna)

INTERVENTIONS:
Drug: Nilotinib (Tasigna) — Patients will be treated with Nilotinib 400 mg two times a day for 6 months.

SUMMARY:
A phase IIa open-label single center pilot study to assess the safety and efficacy of Nilotinib in patients with Scleroderma.

DETAILED DESCRIPTION:
The purpose of this study is to learn how safe and tolerable a medication called Nilotinib (Tasigna) will be for patients diagnosed with Systemic Sclerosis. Systemic Sclerosis (scleroderma) is an autoimmune disease that can involve the skin, the blood vessels, the muscles and other connective tissues, and major organs including the lungs, kidneys, gastrointestinal tract, and heart. The exact cause of this disorder is not known at this time and no drug has been proven to cure scleroderma. Experiments done in animal models and "test-tube" models of fibrosis suggest that Nilotinib may be a useful therapy for scleroderma. Nilotinib is a medication on the market which has been FDA approved for the treatment of a type of leukemia called chronic myelogenous leukemia (CML). It is an oral medication, taken two times a day.

This is a 32 week, open-label, Phase IIa, single center clinical trial. The primary goal of the study is to assess the safety and tolerability of Nilotinib in patients with scleroderma. The secondary goal is to assess how effective Nilotinib is in treating patients with scleroderma. The clinical tests performed such as the Modified Rodnan Skin Score, Pulmonary Function Tests, Echocardiograms, Electrocardiograms, and the blood and skin collected in this study will help determine whether this therapy is safe and effective, and also improve our understanding of scleroderma.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to eighteen years.
2. Clinical diagnosis of diffuse systemic sclerosis by ACR criteria, with a stable modified Rodnan skin score in the one month preceding introduction of oral nilotinib therapy. The modified Rodnan skin score must be greater than or equal to sixteen at screening and initiation of therapy.
3. Disease duration of less than or equal to 3 years as defined by the date of onset of the first non-Raynaud's symptom.
4. Estimated ejection fraction of greater than 50% by echocardiography

Exclusion Criteria:

1. Inability to render informed consent in accordance with institutional guidelines.
2. Disease duration of greater than 3 years.
3. Patients with mixed connective tissue disease or "overlap" (i.e. those who satisfy more than one set of ACR criteria for a rheumatic disease.)
4. Limited scleroderma.
5. Systemic sclerosis-like illness associated with environmental or ingested agents such as toxic rapeseed oil, vinyl chloride, or bleomycin.
6. Ongoing treatment with immunosuppressive therapies including cyclophosphamide, azathioprine, mycophenolic acid, methotrexate, or cyclosporine, or use of those medications within 1 month of trial entry.
7. The use of other anti-fibrotic agents including colchicine, D-penicillamine, minocycline, or Type 1 oral Collagen in the month prior to enrollment.
8. Use in the prior month of corticosteroids at doses exceeding the equivalent of prednisone 10 mg daily. Use of corticosteroid at < 10 mg of prednisone can continue during the course of the study.
9. Concurrent serious medical condition which in the opinion of the investigator makes the patient inappropriate for this study such as uncontrollable CHF, arrhythmia, severe pulmonary or systemic hypertension, severe GI involvement, hepatic impairment, serum creatinine of greater than 2.0, active infection, severe diabetes, unstable atherosclerotic cardiovascular disease, malignancy, HIV, or severe peripheral vascular disease.
10. History of pancreatitis.
11. Prolonged QTc interval defined as a QTc > 450 msec
12. Patients requiring the ongoing use of medications that are antiarrhythmics (including, but not limited to amiodarone, disopyramide, procainamide, quinidine and sotalol) or that prolong the QTc interval (including, but not limited to chloroquine, halofantrine, clarithromycin, haloperidol, methadone, moxifloxacin, bepridil and pimozide) will be excluded.
13. Patients requiring the ongoing use of medications that are potent inhibitors or inducers of CYP3A4.
14. A positive pregnancy test at entry into this study. Men and women with reproductive potential will be required to use effective means of contraception through the course of the study.
15. Participation in another clinical research study involving the evaluation of another investigational drug within ninety days of entry into this study.
16. The presence of severe lung disease as defined by a diffusion capacity of less than 30% of predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spiera, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] Haddon DJ, Wand HE, Jarrell JA, Spiera RF, Utz PJ, Gordon JK, Chung LS. Proteomic Analysis of Sera from Individuals with Diffuse Cutaneous Systemic Sclerosis Reveals a Multianalyte Signature Associated with Clinical Improvement during Imatinib Mesylate Treatment. J Rheumatol. 2017 May;44(5):631-638. doi: 10.3899/jrheum.160833. Epub 2017 Mar 15. PMID 28298564
- [Derived] Gordon JK, Martyanov V, Magro C, Wildman HF, Wood TA, Huang WT, Crow MK, Whitfield ML, Spiera RF. Nilotinib (Tasigna) in the treatment of early diffuse systemic sclerosis: an open-label, pilot clinical trial. Arthritis Res Ther. 2015 Aug 18;17(1):213. doi: 10.1186/s13075-015-0721-3. PMID 26283632

RESULTS

PARTICIPANT FLOW:
Groups:
- Nilotinib 400 mg Twice Daily: Nilotinib (Tasigna): Patients will be treated with Nilotinib 400 mg two times a day for 6 months and could continue treatment for at least 12 months.
Period: Overall Study
Arm/Group | Nilotinib 400 mg Twice Daily
Started | 10
Completed | 7
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib 400 mg Twice Daily
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 8
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 46 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Disease Duration, median (range) [Median (Full Range); unit: years] | 0.7 [0.5 to 1.7]
ANA-positive, n (%) [Count of Participants; unit: Participants] | 9
Anti-Scl 70-positive, n (%) [Count of Participants; unit: Participants] | 3
RNA polymerase III-positive, n (%) [Count of Participants; unit: Participants] | 5
Modified Rodnan Skin Score (MRSS) at baseline [Mean (Standard Deviation); unit: units on a scale] — The Modified Rodnan Skin Score (MRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. In each of these areas, the skin score is evaluated by manual palpation. The skin score is 0 for uninvolved skin, 1 for mild thickening, 2 for moderate thickening, and 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas. The minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease.
  units on a scale | 30.1 (8.2)
Mean change in MRSS in 1 month prior to baseline [Mean (Standard Deviation); unit: units on a scale] — The Modified Rodnan Skin Score (MRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. The skin score is 0 for uninvolved skin through 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas. The minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease. The mean change in MRSS represents the average change in total skin score in 1 month before baseline.
  units on a scale | 2.9 (3.4)
Tendon friction rubs, n (%) [Count of Participants; unit: Participants] | 4
Previous treatment, n (%) [Count of Participants; unit: Participants] | 0
Methotrexate [Count of Participants; unit: Participants] | 2
No immunosuppression [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: 6 Months and 12 months treatment
Measure: Number; unit: Adverse Events
Arm/Group | Nilotinib 400 mg Twice Daily
Number analyzed (Participants) | 7
Adverse Events | 71

2. Secondary Outcome: Improvement of Modified Rodnan Skin Score Reported as a Mean (Units Equals Number of Points)
Description: Efficacy of Nilotinib in patients with systemic sclerosis, as defined by an improvement in the Modified Rodnan Skin Score (MRSS) The Modified Rodnan Skin Score (MRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. The skin score is evaluated by manual palpation in each of these areas. The skin score is 0 for uninvolved skin, 1 for mild thickening, 2 for moderate thickening, and 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas where the minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease.
Time Frame: 6 Months of treatment
Measure: Number; unit: units on a scale
Arm/Group | Nilotinib 400 mg Twice Daily
Number analyzed (Participants) | 7
units on a scale | 4.2

3. Secondary Outcome: Efficacy of Nilotinib in Patients With Systemic Sclerosis, as Defined by an Improvement in the Modified Rodnan Skin Score
Description: Improvement in Modified Rodnan skin score reported as a mean (units equals number of points).
  The Modified Rodnan Skin Score (MRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. In each of these areas, the skin score is evaluated by manual palpation. The skin score is 0 for uninvolved skin, 1 for mild thickening, 2 for moderate thickening, and 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas. The minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease.
Time Frame: 12 months treatment
Measure: Number; unit: units on a scale
Arm/Group | Nilotinib 400 mg Twice Daily
Number analyzed (Participants) | 7
units on a scale | 6.3

ADVERSE EVENTS:
Time Frame: Adverse Event events including Serious Adverse Events were observed during the 12-month treatment period.
Arm/Group | Nilotinib 400 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib 400 mg Twice Daily (N=7)
Syncopal Episode (Cardiac disorders) | 1 — Patient was hospitalized. Medication was held and the patient's evaluation was normal. When the patient followed up and off medication for 3 weeks, baseline was QTc >450 msec and could not restart medication since now met an exclusion criterion.
Coronary Artery Bypass Graft (CABG) Surgery (Vascular disorders) | 1 — Hospitalized for surgery after 3 months treatment. Patient had multiple risk factors for vascular disease and there is possibility that worsening of vascular disease was related to nilotinib use.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nilotinib 400 mg Twice Daily (N=7)
Prolonged QTC (Cardiac disorders) | 6 (9)
Increased AST (Investigations) | 5 (6)
Elevated Total Bilirubin (Investigations) | 5 (6)
Increased ALT (Investigations) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Nausea (Ear and labyrinth disorders) | 2 (2)
Reflux (Gastrointestinal disorders) | 2 (2)
Elevated ESR (Blood and lymphatic system disorders) | 2 (2)
Increased Lipase (Investigations) | 2 (2)
Increased Amylase (Investigations) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Metabolism and nutrition disorders) | 1 (2)
Decreased White Blood Cell Count (Blood and lymphatic system disorders) | 1 (1)
Increased White Blood Cell Count (Blood and lymphatic system disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hospitalization for CABG (Cardiac disorders) | 1 (1)
Allergic Rhinitis (Infections and infestations) | 1 (1)
Cataracts (Eye disorders) | 1 (1)
Conjuctivitis (Eye disorders) | 1 (1)
Eye Disorder (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Interim Bacterial Sinusitis (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Low Inorganic Phosphorus (Metabolism and nutrition disorders) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1)
Ankle Arthiritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Plantar Fascitis (Skin and subcutaneous tissue disorders) | 1 (1)
Calcinosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Concentration Impairment (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes